CLINICAL TRIAL: NCT04987541
Title: The Therapeutic Effect of TBS Stimulation Over Left Dorsolateral Prefrontal Cortex on Emotion Regulation in Autism Spectrum Disorder
Brief Title: The Therapeutic Effect of TBS Stimulation on Emotion Regulation in Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202002498A0
Record Dates: First submitted 2021-07-12; First posted 2021-08-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Participants received the real intervention of TBS (iTBS 600) over the left dorsolateral prefrontal cortex for 4 weeks (5 days/week).
  *iTBS = intermittent theta burst stimulation
  Interventions: Device: intermittent theta burst stimulation
- Sham (Sham Comparator): Participants received the sham intervention of TBS (sham-coil) over the left dorsolateral prefrontal cortex for 4 weeks (5 days/week).
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — stimulatory protocol

SUMMARY:
The investigator would like to investigate the impact of intermittent theta burst stimulation over left dorsolateral prefrontal cortex on emotion regulation in autism spectrum disorder

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum disorder, confirmed by ADOS

Exclusion Criteria:

* Previous or current severe neurological disorder such as epilepsy, visual or hearing impairment
* Previous or current severe systemic disease such as cardiovascular disease, diabetes or infection
* Previous or current severe brain injury
* Implementation of metal materials such as pacemaker or medication pump
* Previous or current severe psychiatric disorders such as schizophrenia, bipolar disorder or substance abuse
* Pregnancy
* Individuals with a significant brain abnormality such as intracranial space occupied lesions
* Individuals with a family history of epilepsy
* Previous febrile seizures
* Current taking antiepileptic drugs
* Concurrent use of medications which increased the risk of seizure attack
* Individuals suffering from sleep deprivation during rTMS procedures
* Skin trauma on application site
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to participate in the study
* Participate another clinical trial within one month

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of total scores of Emotional Dysregulation Inventory | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  Emotional Dysregulation Inventory is a parents' report questionnaire for emotional dysregulation. The score ranges from 0-120. The lower scores stand for better emotional regulation.
Changes of total scores of Aberrant Behavior Checklist | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  ABC is a parents' report questionnaire for aberrant behavior. The lower scores stand for less aberrant behavior.
Changes of total scores of Child Behavior Checklist | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  CBCL is a parents' report questionnaire for behavioral and emotional problems. The lower scores stand for better behavioral and emotional regulation.

SECONDARY OUTCOMES:
Changes of total scores of Social Responsiveness Scale | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  Social Responsiveness Scale can measure the autism clinical severity with the range from 65-260. The lower scores stand for better social responsiveness.
Changes of total scores of Repetitive Behavior Scale-Revised | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  Repetitive Behavior Scale-Revised is a questionnaire that focuses on repetitive behavior. The score ranges from 0-129. The lower scores stand for lower repetitive behavior.
Changes of total scores of Adaptive Behavior Assessment System | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  Adaptive Behavior Assessment System is a parents' report questionnaire for adaptive behavior. The score ranges from 9-171. The higher scores stand for better adaptive behavior.
Changes in accuracy of Frith-Happe animation | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition.
Changes in accuracy of Eyes task | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills.
Changes in accuracy of Wisconsin Card Sorting Test | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  An advanced test for cognitive flexibility. 128 questions in total, the more correct questions stand for better cognitive flexibility.
Changes of total scores of Behavior Rating Inventory of Executive Function | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  Behavior Rating Inventory of Executive Function is a parents' report questionnaire for executive function. The score ranges from 86-258. The lower scores stand for better executive function.
Raven's Progressive Matrices | baseline; post TBS (4 weeks after baseline); One month follow up (4 weeks after post TBS); Two months follow up (8 weeks after post TBS)
  An advanced test for for executive function. 60 questions in total, the more correct questions stand for better executive function.
MRI T1 | baseline; post TBS (4 weeks after baseline)
  Brain structural volumes (cm²)
functional MRI (resting-state/biological motion task) - BOLD signal | baseline; post TBS (4 weeks after baseline)
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI, which reflects the neural activity.
Diffusion Tensor Imaging (DTI) - FA | baseline; post TBS (4 weeks after baseline)
  Fractional anisotropy (FA) is a measurement used in DTI, which reflects the movement of water molecules. FA ranges from 0 to 1, the higher FA value may represent more intact axons.
Electroencephalography | baseline; post TBS (4 weeks after baseline)
  Resting state EEG (alpha power / frontal gamma power)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided